CLINICAL TRIAL: NCT04651569
Title: A Multicentre, Retrospective, Observational Study to Analyse the Efficacy of High Dose Isofosfamide Administered Through Elastomer in Patients With Relapsed/ Refractory Osteosarcoma
Brief Title: An Analysis of the Efficacy of High Dose Isofosfamide Through Elastomer
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera Ospedale Infantile Regina Margherita Sant'Anna (Other)
Responsible Party: Principal Investigator, Prof. Franca Fagioli, Principal Investigator, Azienda Ospedaliera Ospedale Infantile Regina Margherita Sant'Anna
Other Study IDs: HD-IFOel
Record Dates: First submitted 2020-11-25; First posted 2020-12-03 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Osteosarcoma Recurrent
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational study — none, Observational study

SUMMARY:
A multicentre, observational, retrospective study to analyse the efficacy of high dose isofosfamide thorugh elastomer in patients with relapsed/ refractory osteosarcoma

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of high risk relapsed/ refractory osteosarcoma
* Aged <= 40 years at the beginning of treatment
* at least one completed cycle of HD IFO through elastomer (14g/mq) in 14 days
* disease evaluation according to RECIST criteria v.1.1

Exclusion Criteria:

* none

Max Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients with relapsed/ refractory osteosarcom
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | Evaluated during the first 4 months at the end of treatment
  Disease remission or disease progression
growth modulation index - GMI | Evaluation to be recorded at each disease assessment through imaging (PET/CT/MRI)
  ratio of time to progression (TTP) with nth line of therapy (TTPn) to the most recent prior line of therapy (TTPn-1)
toxicity according to CTCAE v.5.0 | Evaluation to be recorded at each disease assessment through imaging (PET/CT/MRI)
  Disease evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Celeste Cagnazzo, PhD, Study Chair — A.O.U. Città della Salute e della Scienza
Locations (5):
- Italy (5):
  - Istituto Ortopedico Rizzoli, Bologna
  - Azienda Ospedaliero Universitaria Meyer, Florence
  - IRCCS Istituto Nazionale dei Tumori - S.C. Pediatria, Milan
  - Regina Elena National Cancer Institute IRCCS, Roma
  - OIRM - AOU Città della Salute e della Scienza di Torino, Torino

IPD SHARING:
Plan to Share IPD: No